CLINICAL TRIAL: NCT02845596
Title: Unrelated Donor Transplant Versus Immune Therapy in Pediatric Severe Aplastic Anemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michael Pulsipher (Other)
Responsible Party: Sponsor-Investigator, Michael Pulsipher, Principal Investigator, Pediatric Transplantation & Cellular Therapy Consortium
Organization: Pediatric Transplantation & Cellular Therapy Consortium (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TransIT NMD 1601
Record Dates: First submitted 2016-05-09; First posted 2016-07-27 (Estimated); Last update posted 2025-05-11 (Actual); Status verified 2024-04

CONDITIONS: Severe Aplastic Anemia
MeSH Terms: conditions — Anemia, Aplastic | interventions — Cyclosporine; Antilymphocyte Serum; thymoglobulin; Methotrexate; fludarabine; Cyclophosphamide; Whole-Body Irradiation; Immunosuppression Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immunosuppressive Therapy (Active Comparator): Patient will receive standard immunosuppressive therapy combination of drugs: horse anti-thymocyte globulin (ATG) and cyclosporine.
  Interventions: Drug: cyclosporine; Drug: horse anti-thymocyte globulin (ATG); Procedure: Immunosuppressive Therapy (IST)
- Matched Unrelated Stem Cell Transplant (Active Comparator): Patient will under go matched unrelated donor transplant of hematopoietic stem cells as their therapy using fludarabine, cyclophosphamide, rabbit anti-thymocyte globulin (ATG), and low-dose total body irradiation (TBI) as preparative regimen and cyclosporine and methotrexate for graft versus host disease (GVHD) prevention.
  Interventions: Drug: cyclosporine; Procedure: Matched Unrelated Donor Hematopoietic Stem Cell Transplant; Drug: rabbit anti-thymocyte globulin (ATG); Drug: methotrexate; Drug: fludarabine; Drug: cyclophosphamide; Radiation: low-dose total body irradiation (TBI)

INTERVENTIONS:
Drug: cyclosporine — cyclosporine
Procedure: Matched Unrelated Donor Hematopoietic Stem Cell Transplant — Matched Unrelated Donor (MUD) Hematopoietic Stem Cell Transplantation (HSCT)
  Arms: Matched Unrelated Stem Cell Transplant
Drug: horse anti-thymocyte globulin (ATG) — horse anti-thymocyte globulin (ATG)
  Other Names: ATGAM
  Arms: Immunosuppressive Therapy
Drug: rabbit anti-thymocyte globulin (ATG) — rabbit anti-thymocyte globulin (ATG)
  Other Names: Thymoglobulin
  Arms: Matched Unrelated Stem Cell Transplant
Drug: methotrexate — methotrexate
  Arms: Matched Unrelated Stem Cell Transplant
Drug: fludarabine — fludarabine
  Arms: Matched Unrelated Stem Cell Transplant
Drug: cyclophosphamide — cyclophosphamide
  Arms: Matched Unrelated Stem Cell Transplant
Radiation: low-dose total body irradiation (TBI) — low-dose total body irradiation (TBI)
  Arms: Matched Unrelated Stem Cell Transplant
Procedure: Immunosuppressive Therapy (IST) — Immunosuppressive Therapy (IST)
  Arms: Immunosuppressive Therapy

SUMMARY:
The purpose of this study is to determine the feasibility of comparing outcomes of patients treated de novo with immunosuppressive therapy (IST) versus matched unrelated donor (MUD) hematopoietic stem cell transplant (HSCT) for pediatric acquired severe aplastic anemia.

DETAILED DESCRIPTION:
A major challenge in treating pediatric Severe Aplastic Anemia (SAA) is the determination of best primary therapy for patients who lack a fully matched related donor for HSCT. Good survival outcomes have been seen with IST, but initial and late failures, CSA dependence, persistent cytopenias and secondary Myelodysplastic Syndrome (MDS) / Acute Myeloid Leukemia (AML) in a portion of patients leave considerable room for improvement. MUD HSCT survival in SAA has markedly improved, but a direct comparison of this approach with IST is necessary to determine whether this approach is feasible and will lead to better Event Free Survival. This trial will address the feasibility of randomization, test whether patients can be evaluated in a timely fashion and safely begin therapy with MUD HSCT or IST, and give a preliminary assessment of the safety of up-front MUD HSCT. If successful, this trial will lead to a future prospective trial comparing directly IST to MUD HSCT in this disease.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of idiopathic SAA, defined as:

   * Bone marrow cellularity <25%, or <30% hematopoietic cells.
   * Two out of three of the following (in peripheral blood): neutrophils <0.5 x109/L, platelets <20 x109/L, reticulocyte count <60 x109/L with hemoglobin <8g/dL.
2. Age ≤25 years old.
3. No suitable fully matched related donor available (minimum 6/6 match for Human Leukocyte antigen (HLA) -A and B at intermediate or high resolution and DRB1 at high resolution using DNA based typing).
4. At least two unrelated donors noted on National Marrow Donor Program (NMDP) search who are well matched (9/10 or 10/10 for HLA-A, B, C, DRB1, and DQB1 using high resolution).
5. Signed informed consent for the randomized trial by patient and/or legal guardian.
6. Adequate organ function defined as in the judgment of the investigator, there is not irreversible organ damage that would preclude the patient from meeting the organ function inclusion criteria for HSCT listed in section 2.3.4 by the intended time of HSCT (6-8 weeks after randomization) or preclude patients from receiving horse ATG.

Exclusion Criteria:

1. Inherited bone marrow failure syndromes (IBMFS). The diagnosis of Fanconi anemia must be excluded by diepoxybutane (DEB) or equivalent testing on peripheral blood or marrow. Telomere length testing should be sent on all patients to exclude Dyskeratosis congenita, but if results are delayed or unavailable and there are no clinical manifestations of DC, patients may enroll. If patients have clinical characteristics suspicious for Shwachman Diamond syndrome, this syndrome must be excluded by pancreatic isoamylase testing or gene mutation analysis. Note: pancreatic isoamylase testing is not accurate in children less than 3 years.
2. Clonal cytogenetic abnormalities or fluorescence In Situ Hybridization (FISH) pattern consistent with pre-myelodysplastic syndrome (pre-MDS) or MDS on marrow examination (see section 4.2.3.1 for details of the required MDS FISH panel).
3. Known severe allergy to horse ATG.
4. Prior allogeneic stem cell transplant.
5. Prior solid organ transplant.
6. Infection with human immunodeficiency virus (HIV).
7. Active Hepatitis B or C. This should be excluded in patients where there is clinical suspicion of hepatitis (e.g. elevated LFTs).
8. Female patients who are pregnant or breast-feeding.
9. Prior malignancies except resected basal cell carcinoma or treated cervical carcinoma in situ.

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-08; Primary Completion 2020-11-03 (Actual); Study Completion 2023-07-19 (Actual)

PRIMARY OUTCOMES:
Percentage of patients randomized to HSCT that actually complete HSCT | 4 years
  Feasibility of comparing outcomes of patients treated de novo with IST versus matched unrelated donor HSCT for pediatric acquired severe aplastic anemia as defined by percentage of patients randomized to HSCT that actually complete HSCT.

SECONDARY OUTCOMES:
Time from screening consent to randomization | 4 years
  To measure the time from screening consent and randomization of patients to initiation of the preparative regimen of those randomized to HSCT.
Number of patients that fail to receive their primary assigned therapy (HSCT or IST). | 4 years
  Number of patients fail to receive their primary assigned therapy (HSCT or IST).
Reasons why patients fail to receive their primary assigned therapy (HSCT or IST). | 4 years
  Reasons why patients fail to receive their primary assigned therapy (HSCT or IST).
Treatment-related mortality at one year from randomization in both arms | 1 Year
  Number of deaths that are treatment related
Overall Survival at one year from randomization in both arms | 1 Year
  percentage of enrolled patients living at 1 year post randomization
Time from randomization to neutrophil recovery in both arms | 4 years
  Time from randomization to neutrophil recovery in both arms
Time from randomization to platelet recovery in both arms | 4 years
  Time from randomization to platelet recovery in both arms
Time from randomization to red blood cell recovery in both arms | 4 years
  Time from randomization to red blood cell recovery in both arms
Time from randomization to cessation of immune suppression recovery in both arms | 4 years
  Time from randomization to cessation of immune suppression recovery in both arms
Rates of primary and secondary graft rejection in the MUD HSCT arm | 4 years
  Rates of primary and secondary graft rejection in the MUD HSCT arm
Rates of grade II-IV and III-IV acute GVHD, and extensive chronic GVHD in the MUD HSCT arm | 4 years
  Rates of grade II-IV and III-IV acute GVHD, and extensive chronic GVHD in the MUD HSCT arm
Rates of IST response | 4 years
  Rates of IST response
Rates of IST relapse | 4 years
  Rates of IST relapse
Rates of secondary MDS or AML in both treatment arms. | 4 years
  Rates of secondary MDS or AML in both treatment arms.
Rates of other secondary malignancies in both treatment arms. | 4 years
  Rates of other secondary malignancies in both treatment arms.
Development of symptomatic PNH in both treatment arms. | 4 years
  Development of symptomatic PNH in both treatment arms.
Incidence of significant infection in both treatment arms | 4 years
  Incidence of significant infection in both treatment arms
Time to immune reconstitution in the HSCT arm | 4 years
  Time to immune reconstitution in the HSCT arm

CONTACTS AND LOCATIONS:
Overall Officials: Michael Pulsipher, MD, Study Chair — Children's Hospital Los Angeles; David A Williams, MD, Study Chair — Boston's Childrens Hospital
Locations (13):
- United States (13):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Stanford Lucile Packard Children's Hospital, Palo Alto, California
  - UCSF, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Boston Children's Hospital, Boston, Massachusetts
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Cohen Children's Medical Center, Queens, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided